CLINICAL TRIAL: NCT00150917
Title: A Randomized Controlled Trial of a Group Intervention for Women With a Family History of Breast Cancer
Brief Title: RCT of a Group Intervention for Women With a Family History of Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Breast Cancer Research Alliance (Other); Canadian Cancer Trials Group (Network)
Responsible Party: Dr. Mary Jane Esplen, University Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UHN02-0603-E; CBCRA 015445
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2006-12

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; Genetics; Psychotherapy; Group counselling; Randomized control trial; Risk counselling; Women's mental health; Familial breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Supportive-Expressive Group Therapy

SUMMARY:
One in 10 Canadian women will be diagnosed with breast cancer (BC) and approximately 5% of all BC is believed to be hereditary. Women with a family history experience high levels of perceived risk for developing BC. Elevated risk perceptions for BC have been associated with psychological distress, which, in turn, can interfere with screening adherence. In our completed CBCRI-funded study, we developed and standardized a group intervention designed to address the psychological issues associated with having a family history of BC. Results demonstrated that the intervention led to significant improvement in levels of anxiety and depression, improved BC risk factors/genetics knowledge and was associated with optimal screening behavior. The proposed study will rigorously test the group intervention in comparison to standard risk counselling in a sample of 150 women recruited from Familial BC clinics in Toronto. The interventions will be examined for their impact on a) psychological functioning, b) BC risk/genetic knowledge and c) screening behaviors.

DETAILED DESCRIPTION:
Keywords: Breast cancer, genetics, psychotherapy, group counselling, randomized control trial, risk counselling, women's mental health, familial breast cancer.

One in 10 Canadian women will be diagnosed with breast cancer (BC) and approximately 5% of all BC is believed to be hereditary. Women with a family history of BC experience high levels of perceived risk and vulnerability for developing BC. Elevated risk perceptions for BC are difficult to modify and have been associated with psychological distress that, in turn, can interfere with screening adherence. The specific objectives of the current randomized trial are to determine the effects of a supportive-expressive group intervention on a) psychosocial functioning (using standardized instruments), b) BC risk/genetic knowledge and c) screening behaviors in women with a family history of breast cancer receiving standard genetic risk counseling. Preliminary data will be collected to examine the cost effectiveness of the intervention.

The study is being conducted in the following University of Toronto affiliated teaching hospitals: Mount Sinai Hospital; Preventive Oncology Program, Sunnybrook and Women's College Health Sciences; Toronto Sunnybrook Regional Cancer Centre; University Health Network; North York General Hospital; Credit Valley Hospital. A total of 150 women with a family history of BC will be randomized in a ratio of 2 to 1 to participate in an 8 weekly/ 4 monthly support group or to a control arm that receives educational materials.

The study has been funded by the Canadian Breast Cancer Research Initiative (CBCRI) of the National Cancer Institute of Canada since 2001. To date 66 women have been enrolled in the study and we anticipate a total of 90 women will be enrolled by the end of the current funding year in June 2004. At this rate it is expected that recruitment will be completed in June 2005, the last intervention groups will be completed by January 2006 and that analysis of the final study results will be completed by June 2006. Analysis of baseline data will begin in September 2005 once the last study groups have been initiated and a manuscript reporting the final results will be prepared by June 2006. Two years of funding is requested for these activities.

Significance: Technological advances in molecular biology and genetics are occurring rapidly. Our proposed research has direct relevance for advancing knowledge on the communication and provision of risk/genetic information to individuals with a family history of BC and has both direct and indirect relevance to individuals at all stages of cancer. Improved counselling techniques for those with a family history may impact on the prevention and management of BC through improved surveillance and preventive techniques, enhanced psychosocial functioning and wellbeing through increased psychological resilience. In addition, effective risk counselling interventions may facilitate the understanding of and decision-making around genetic testing, and the adjustment to a cancer diagnosis, should these women with family histories later develop the disease.

ELIGIBILITY:
Inclusion Criteria:

* at least one 1st-degree relative with Breast Cancer
* age 18-70 years
* live within one hour of downtown Toronto
* score higher than 15 in Breast Cancer Anxiety Scale (BCAS)

Exclusion Criteria:

* Carrier status for genetic mutation (i.e. BRCA1) known
* Previous diagnosis of breast cancer or other malignancy (other than non-melanoma skin cancer)
* History of major psychiatric disorder, such as schizophrenia, active psychosis, untreated major depression, as defined in the DSM IV and obtained through a semi-structured psychiatric interview
* Failure to provide informed consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2001-07; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Psychosocial functioning (using standardized instruments) | 1 year
Breast Cancer risk/genetic knowledge | 1 year
Screening behaviors | 1 year

SECONDARY OUTCOMES:
Post Traumatic Growth | 1 year
Cost effectiveness | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Esplen, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada